CLINICAL TRIAL: NCT01142531
Title: Effects of Bronchodilation on CT Parameters Reflecting Airways Remodelling, and Pulmonary Emphysema Extent: Comparisons Between CT Scans Obtained Before and After Bronchodilation and Relationships With Pulmonary Function Tests.
Brief Title: Effects of Bronchodilation on Computed Tomography (CT) Parameters Reflecting Airways Remodelling, and Pulmonary Emphysema Extent.
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Collaborators: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Maxime HACKX, Maxime HACKX, MD, Erasme University Hospital
Other Study IDs: AK/10-02-13/3862
Record Dates: First submitted 2010-04-12; First posted 2010-06-11 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: COPD; CT; Bronchodilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD: COPD patients aged 40 or more, with a smoking history of > 10 PY and a post-bronchodilator FEV1/VC < 0.7 will be included. Exclusion criteria are: COPD exacerbation or respiratory infection in the 4 weeks before the begin of the study, concomitant pulmonary disease (tuberculosis, significant bronchiectasis, lung cancer), pulmonary resection, active malignancy or malignancy of any organ system within the past 5y.
  Interventions: Radiation: Chest CT scan

INTERVENTIONS:
Radiation: Chest CT scan — Supine CT scan after full inspiration. Acquisition parameters: (Topogram 35 mA 120 kV 512 mm length)
  * 90 quality ref mAs with care-dose ON
  * 120 kV
  * Pitch 1.4
  * Rotation time 0.33 s
  * Acquired images 64 x 0.6 mm

SUMMARY:
CT studies considering bronchial dimensions in chronic obstructive pulmonary disease (COPD) were conducted without control of bronchodilation. Some data however suggest that total lung capacity (CT scan is performed after full inspiration) is increased in individuals affected by chronic or spontaneous bronchoconstriction and may decrease after bronchodilatation. Furthermore, no study has assessed the effect of bronchodilation on CT scans parameters reflecting airway remodelling and emphysema extent in COPD patients.

This is a prospective study whose purpose is to assess the effect of bronchodilation on lung CT scan and pulmonary function testing (PFT) in COPD patients.

DETAILED DESCRIPTION:
Patients : COPD patients aged 40 years or more, with a smoking history of > 10 pack-years (PY) and a post-bronchodilator forced expiratory volume in one second to vital capacity ratio (FEV1/VC) < 0.7 will be included. Exclusion criteria are: COPD exacerbation or respiratory infection in the 4 weeks before the begin of the study, concomitant pulmonary disease (tuberculosis, significant bronchiectasis, lung cancer), pulmonary resection, active malignancy or malignancy of any organ system within the past 5 years.

Procedures:

At Visit 1, after obtaining the written informed consent of the patient, medical history, smoking status and patient's treatment will be collected. They will be asked to discontinue bronchodilator therapies as follows, such that pulmonary function tests (PFT) and CT scan will be initially evaluated in a medication wash-out period at Visit 2:

* Short acting a2 agonists and anticholinergics: 8 wash-out
* Long acting a2 agonists: 12h wash-out
* Long acting anticholinergics: 48h wash-out
* Theophylline preparations: 48h wash-out
* Antileucotrienes: 48h wash-out

At visit 2, PFT will be performed, including vital capacity (VC), forced vital capacity (FVC), functional residual capacity (FRC), total lung capacity (TLC), residual volume (RV), forced expiratory volume in one second (FEV1), diffusion lung capacity for carbon monoxide (DLCO), and alveolar volume (VA) measurements (either in absolute values and percentage of predicted values). A first CT scan will be performed using the following technique:

* Supine CT scan after full inspiration.
* Acquisition parameters: (Topogram 35 mA 120 kV 512 mm length) 90 quality ref mAs with care-dose ON 120 kV Pitch 1.4 Rotation time 0.33 s Acquired images 64 x 0.6 mm
* Reconstructions parameters:

B60f 1mm-thick every 0.7 mm B20f 1mm-thick every 10.0 mm B35f 1mm-thick every 0.7 mm B60f 5mm-thick every 5.0 mm B35f 5mm-thick every 5.0 mm

After the initial PFT and CT scan, the patient will receive 80 µg of ipratropium bromide(= 4X20µg Atrovent, via Metered-Dose Inhaler + spacer, 30 seconds between each dose) and 60 minutes later, 400 µg salbutamol (=4X100 µg Ventolin).

A second PFT will be performed 30 min after salbutamol inhalation, followed by a second CT Scan.

Data analysis:

* Emphysema index: from B20f reconstructions, calculation of RA960 using Pulmo CT software.
* Airway index: from B60f reconstructions (1mm-thick every 0.7 mm), calculations of luminal area and wall area for several bronchi.

Statistical analyses : Comparisons of CT parameters values or derived values (for example : wall area to airway area ratio) reflecting emphysema and airways remodelling, before and after bronchodilation. Correlations with PFT values and derived values.

ELIGIBILITY:
Inclusion Criteria:

* age 40 or more
* Smoking history > 10 pack-years
* post bronchodilator FEV1/VC < 0.7

Exclusion Criteria:

* COPD exacerbation or infection in the 4 weeks before the study
* Concomitant pulmonary disease (tuberculosis, significant bronchiectasis, lung cancer)
* pulmonary resection
* active malignancy or malignancy of any organ system within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients aged 40 or more, with a smoking history of > 10 PY and a post-bronchodilator FEV1/VC < 0.7 will be included. Exclusion criteria are: COPD exacerbation or respiratory infection in the 4 weeks before the begin of the study, concomitant pulmonary disease (tuberculosis, significant bronchiectasis, lung cancer), pulmonary resection, active malignancy or malignancy of any organ system within the past 5y.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Results of CT Thorax parameters reflecting emphysema airway remodelling | 4 hours
  Data analysis:
  * Emphysema index: from B20f reconstructions, calculation of RA960 using Pulmo CT software.
  * Airway index: from B60f reconstructions (1mm-thick every 0.7 mm), calculations of luminal area and wall area for several bronchi.

SECONDARY OUTCOMES:
Results of pulmonary function tests | 4 hours
  Pulmonary function tests will be performed before and after bronchodilation:
  vital capacity (VC), forced vital capacity (FVC), functional residual capacity (FRC), total lung capacity (TLC), residual volume (RV), forced expiratory volume in one second (FEV1), diffusion lung capacity for carbon monoxide

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alain GEVENOIS, MD, PhD, Study Director — Erasme University Hospital
Locations (1):
- C.H.U Saint-Pierre, Brussels, Belgium

REFERENCES:
- [Background] Nakano Y, Muro S, Sakai H, Hirai T, Chin K, Tsukino M, Nishimura K, Itoh H, Pare PD, Hogg JC, Mishima M. Computed tomographic measurements of airway dimensions and emphysema in smokers. Correlation with lung function. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1102-8. doi: 10.1164/ajrccm.162.3.9907120. PMID 10988137
- [Background] Hasegawa M, Nasuhara Y, Onodera Y, Makita H, Nagai K, Fuke S, Ito Y, Betsuyaku T, Nishimura M. Airflow limitation and airway dimensions in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1309-15. doi: 10.1164/rccm.200601-037OC. Epub 2006 Mar 23. PMID 16556695
- [Background] Patel BD, Coxson HO, Pillai SG, Agusti AG, Calverley PM, Donner CF, Make BJ, Muller NL, Rennard SI, Vestbo J, Wouters EF, Hiorns MP, Nakano Y, Camp PG, Nasute Fauerbach PV, Screaton NJ, Campbell EJ, Anderson WH, Pare PD, Levy RD, Lake SL, Silverman EK, Lomas DA; International COPD Genetics Network. Airway wall thickening and emphysema show independent familial aggregation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Sep 1;178(5):500-5. doi: 10.1164/rccm.200801-059OC. Epub 2008 Jun 19. PMID 18565956
- [Background] Duranti R, Filippelli M, Bianchi R, Romagnoli I, Pellegrino R, Brusasco V, Scano G. Inspiratory capacity and decrease in lung hyperinflation with albuterol in COPD. Chest. 2002 Dec;122(6):2009-14. doi: 10.1378/chest.122.6.2009. PMID 12475840
- [Background] Pellegrino R, Brusasco V. On the causes of lung hyperinflation during bronchoconstriction. Eur Respir J. 1997 Feb;10(2):468-75. doi: 10.1183/09031936.97.10020468. PMID 9042651
- [Background] Stanescu DC, Rodenstein D, Cauberghs M, Van de Woestijne KP. Failure of body plethysmography in bronchial asthma. J Appl Physiol Respir Environ Exerc Physiol. 1982 Apr;52(4):939-48. doi: 10.1152/jappl.1982.52.4.939. PMID 7085427
- [Background] Berger P, Perot V, Desbarats P, Tunon-de-Lara JM, Marthan R, Laurent F. Airway wall thickness in cigarette smokers: quantitative thin-section CT assessment. Radiology. 2005 Jun;235(3):1055-64. doi: 10.1148/radiol.2353040121. Epub 2005 Apr 15. PMID 15833982
- [Background] Orlandi I, Moroni C, Camiciottoli G, Bartolucci M, Pistolesi M, Villari N, Mascalchi M. Chronic obstructive pulmonary disease: thin-section CT measurement of airway wall thickness and lung attenuation. Radiology. 2005 Feb;234(2):604-10. doi: 10.1148/radiol.2342040013. PMID 15671010
- [Derived] Hackx M, Gyssels E, Severo Garcia T, De Meulder I, Alard S, Bruyneel M, Van Muylem A, Ninane V, Gevenois PA. Chronic Obstructive Pulmonary Disease: CT Quantification of Airway Dimensions, Numbers of Airways to Measure, and Effect of Bronchodilation. Radiology. 2015 Dec;277(3):853-62. doi: 10.1148/radiol.2015140949. Epub 2015 May 19. PMID 25989594